CLINICAL TRIAL: NCT06523114
Title: Transcatheter Arterial Embolization for Relief of Chronic Musculoskeletal Elbow and Foot Plantar Pain Refractory to Conservative Treatment
Brief Title: Transcatheter Arterial Embolization for Elbow and Foot Plantar Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Collaborators: Dongkook Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Woosun Choi, Associate Professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2110-003-449
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Elbow Tendinitis; Elbow Tendinopathy; Epicondylitis of the Elbow; Epicondylitis, Lateral; Plantar Fascitis; Embolization
MeSH Terms: conditions — Elbow Tendinopathy; Tennis Elbow

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lateral epicondylitis and plantar fascitis group (Experimental): Among patients with lateral epicondylitis or plantar fascitis, pain refractory to at least 6 months of physician directed conservative therapy
  Interventions: Device: Transcatheter Arterial Embolization

INTERVENTIONS:
Device: Transcatheter Arterial Embolization — After accessing the common femoral artery or radial artery, embolization is performed using embolic material after confirming abnormal blood vessel abnormalities, lesion hypervascularity, and lesion enhancement findings.

SUMMARY:
This is a prospective single arm study in which patients with moderate to severe chronic elbow or foot plantar pain, in the setting of lateral epicondylitis or plantar fascitis refractory to conservative treatment, will be enrolled.

The primary aim of this study is to estimate the effectiveness and safety of transcatheter arterial embolization (TAE) for changes in elbow or plantar pain with 6 and 12-month follow-up.

DETAILED DESCRIPTION:
This is a prospective single arm, single center study at Chung-Ang University Hospital. Patients with moderate to severe elbow or foot pain, and pain refractory to at least 6 months of physician directed conservative therapy (oral analgesic, physical therapy or local injection treatment) will be eligible for enrollment.

Transcatheter arterial embolization (TAE) is performed after receiving informed consent, and imipenem is used as an embolic material to embolize the target lesion. After the procedure, evaluate the VAS score and limitation of range of motion (LOM) of the joint area.

Follow-up at 1, 3, 6 and 12 months after embolization, and changes of VAS score and LOM are checked.

ELIGIBILITY:
Inclusion Criteria:

* Patients who voluntarily signed a written consent form after receiving an explanation of the purpose, method, and effects of this clinical trial
* Patients who have had pain in the relevant area for more than 6 months and have a history of receiving physical therapy, analgesic anti-inflammatory medication, or local injection treatment
* Patients in whom hypervascularization was confirmed in the relevant area through imaging results (US, CT, MRI) evaluating the cause of pain.

Exclusion Criteria:

* Patients are pregnant or breastfeeding
* Local infection in the painful area
* Patients have a bleeding disease

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale Pain (VAS) Score | 1,3,6,12 month
  At 1 week, 1 month, 3 months, 6 months, and 12 months after the procedure, the degree of pain (visual analog scale pain, 10 points for maximum pain, 0 points for no pain) is assessed through an outpatient visit or by phone.

SECONDARY OUTCOMES:
Adverse Events | 1,3,6,12 month
  Compare the safety of TAE by recording adverse events at 1 month, 3 months, 6 months, and 12 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Woosun Choi, MD. Ph D., Study Director — Associate Professor
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea